CLINICAL TRIAL: NCT06051864
Title: Effectiveness of Electrical Vestibular Nerve Stimulation in the Management of Depression
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) As a Treatment for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: NRI Institute of Medical Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMS001
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active VeNS (Active Comparator): The active device utilizes a technology termed vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Modius Mood Active Device
- Sham VeNS (Placebo Comparator): The sham device looks identical to the active device and interacts with the app in a similar manner to the active device. It will apply some stimulation to a user for a limited period of time (30 seconds), before tapering down to zero over a further 20 seconds, thus creating the impression of an active device. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Modius Mood Active Device — Battery powered non-invasive neurostimulation device
  Arms: Active VeNS
Device: Sham Device — Placebo comparator sham device (no active stimulation)
  Arms: Sham VeNS

SUMMARY:
Trial title: Effectiveness of Electrical Vestibular Nerve Stimulation in the Management of Depression

The aim of this study: To better evaluate the efficacy of non-invasive electrical vestibular nerve stimulation (VeNS) as a method of treating Depression, as compared to a sham control.

Allocation: Randomized to either active device or control device usage.

Endpoint classification: Efficacy Study Intervention Model: Parallel Assignment in 1:1 active to control allocation

Sample size: The aim is to recruit a total of up to 60 participants. The study will last 12 weeks in total for each subject.

DETAILED DESCRIPTION:
This double blind randomized controlled trial will enroll up to 60 subjects and will be conducted at the NRI Institute of Medical Sciences. The study will be randomized for a 8-week period with a 1:1 active to sham device allocation. Each participant will complete 5 stimulation sessions per week under the supervision of a researcher at the Department of Physiology. Each session will be 30 minutes on the day of usage. The scheduled study events are to be undertaken at the following timepoints:

* Baseline: Study Visit 1 (0-week timepoint for enrolment)
* Study Visit 2 (2-week timepoint)
* Study Visit 3 (4-week timepoint)
* Study Visit 4 (6-week timepoint)
* End of Study: Study Visit 5 (8-week timepoint)
* Post-intervention follow-up at 4 weeks (12-week timepoint)

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Male or female, age ≥ 18 years and ≤ 80 years at the time of signing informed consent
* PHQ-9 score of >/=10 at screening
* On anti-depressant medication to treat depression (participant must only be on one Selective Serotonin or Norepinephrine Reuptake Inhibitor (SSRI/SNRI) for at least 1 year prior to baseline visit, and no longer than 5 years
* Stable dose of anti-depressant (SSRI/SNRI) medication to treat depression, 3 months prior to baseline appointment
* Stable medication regime for at least 4 weeks prior to the baseline visit
* Can speak / read Hindi / English
* Ability and willingness to complete all study visits and procedures; in particular an agreement to engage with trying to use the device per the study protocol
* Ability and willingness to adhere to 30 minutes usage of the device at 5 days per week for the duration of the trial at clinic
* Agree not to undergo any extreme lifestyle changes during the duration of the study that could impact sleep e.g. dietary or exercise changes

Exclusion Criteria:

* Patient Health Questionnaire-9 (PHQ-9) score of <10 at screening
* Risk of persistent self-harm or suicide
* Diagnosis or history of bipolar disorder
* History of a current psychotic disorder such as schizophrenia or other non-mood disorder psychosis
* Diagnosis of substance use disorder or dependence
* Use of recreational drugs (e.g nalgesics, depressants, stimulants, and hallucinogens). Subject can enrol after a washout period of 30 days
* History of diagnosed cognitive impairment / disorder such as delirium or dementia
* Previous diagnosis of a chronic viral infection, for example hepatitis or HIV.
* History of stroke or head injury requiring intensive care or neurosurgery
* Presence of permanently implanted battery-powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator, etc.)
* History of epilepsy
* History of severe tinnitus or vertigo
* History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.
* History or presence of malignancy within the last year (except basal and squamous cell skin cancer and in-situ carcinomas)
* History of vestibular dysfunction or another inner ear disease
* Regular use (more than twice a month) of antihistamine medication within the last 6 months
* A diagnosis of myelofibrosis or myelodysplastic syndrome
* Diagnosis of active migraines
* Previous use of Modius device or any VeNS device
* Participation in other clinical trials sponsored by Neurovalens
* Any other medical condition, or medication use, that in the opinion of the PI is likely to make the subject refractory to VeNS.
* Failure to use device daily during trial participation (no more than 14 consecutive days usage drop without reasonable explanation)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-12-03 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of the Modius Mood device, relative to the sham control group, in reducing the severity of depression at 8 weeks | 8 weeks
  Change in the Beck's Depression Inventory (BDI) score from baseline to 8 weeks between the active and control group.

SECONDARY OUTCOMES:
To evaluate the ability of the Modius Mood device, relative to the sham control group, in reducing the severity of depression at 2, 4 and 6 weeks | 8 weeks
  Change in the Beck's Depression Inventory (BDI) score at additional timepoints (2, 4, and 6 weeks) between the active and control group.
To evaluate the impact of the Modius Mood device, relative to the control group, on anxiety at 4 weeks and 8 weeks | 8 weeks
  Change in the Generalized Anxiety Disorder Assessment (GAD-7) score from baseline to 4 weeks and 8 weeks between the active and control group.
To evaluate the impact of the Modius Mood device, relative to the control group, on insomnia at 4 weeks and 8 weeks | 8 weeks
  Change in the Insomnia Severity Index (ISI) score from baseline to 4 weeks and 8 weeks between the active and control group.
To evaluate the effect of the Modius Mood, relative to control group, on quality of life at 4 weeks and 8 weeks | 8 weeks
  Change in the Quality of Life (EQ-5D-5L) score from baseline to 4 weeks and 8 weeks between the active and control group

OTHER OUTCOMES:
To evaluate the safety of the Modius Mood device, relative to control group, in terms of the occurrence of adverse events for the duration of the study | 8 weeks
  An evaluation of the safety of the Modius Mood device will be quantified by the occurrence in adverse events between the active and control group during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Sai Sailesh Kumar Goothy, Principal Investigator — NRI Institute of Medical Sciences
Locations (1):
- NRI Institute of Medical Sciences, Visakhapatnam, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided